CLINICAL TRIAL: NCT03969290
Title: Clinical Performance of Two Daily Disposable Contact Lenses - Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-P001
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Refractive Errors
Keywords: Contact lens; Vision correction; Visual acuity; Daily disposable contact lens
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: Contralateral
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Experimental): Verofilcon A contact lens in the right eye (OD), with etafilcon A contact lens in the left eye (OS), as randomized. Lenses will be worn for one day, approximately 8 hours.
  Interventions: Device: Verofilcon A contact lenses; Device: Etafilcon A contact lenses
- Sequence 2 (Active Comparator): Etafilcon A contact lens in the right eye (OD), with verofilcon A contact lens in the left eye (OS), as randomized. Lenses will be worn for one day, approximately 8 hours.
  Interventions: Device: Verofilcon A contact lenses; Device: Etafilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Daily disposable silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Other Names: Precision1™
Device: Etafilcon A contact lenses — Daily disposable contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia)
  Other Names: Acuvue® Moist

SUMMARY:
The purpose of this study is to evaluate end of day (EOD) visual acuity (VA) at distance when wearing Precision1™ contact lenses compared to Acuvue® Moist contact lenses.

DETAILED DESCRIPTION:
The expected duration of subject participation in the study is 1-8 days, with 3 scheduled visits (Screening, Dispense, Exit).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an approved Informed Consent form
* Successful wear of spherical soft contact lenses for distance correction in both eyes during the past 3 months for a minimum of 5 days per week and 8 hours per day
* Best corrected VA of logMAR 0.10 or better in each eye
* Willing to discontinue artificial tears and rewetting drops during the study
* Able to wear contact lenses within the protocol-specified sphere power range
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, or abnormality or disease that contraindicates contact lens wear, as determined by the Investigator
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator
* History of ocular or intraocular surgery, including refractive surgery, and/or irregular cornea
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment
* Previous 3 years or current wearers of Acuvue Moist or DAILIES TOTAL1® contact lenses
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
End of day (EOD) visual acuity at distance | Day 1, after 8 hours of wear
  Visual acuity (VA) will be measured in "logarithm of the minimum angle of resolution" (logMAR). A lower logMAR value indicates better visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (1):
- Alcon Investigative Site, Jena, Germany

IPD SHARING:
Plan to Share IPD: No